CLINICAL TRIAL: NCT02072577
Title: Effect of Educational Video in the Student's Knowledge About Oral Hygiene of Patients Undergoing Chemotherapy
Brief Title: Effect of Educational Video in the Student's Knowledge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Emilia Campos de Carvalho, Full professor, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 01686312700005393
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2012-05

CONDITIONS: Students of Undergraduate School of Nursing
Keywords: Nursing care, oral health, educational video, oral hygiene.
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Knowledge (Experimental): Educational video.
  Interventions: Behavioral: Video

INTERVENTIONS:
Behavioral: Video — The student watched the video prepared individually in the ward where they were interned.
  After this step, the student demonstrated again the procedure for oral hygiene.
  At this point the researcher also observed the sequence, movements and technical procedures used to analyze the steps of oral hygiene, using the same instrument for such employee initially.

SUMMARY:
Supervise dental conditions and teach the procedure of oral hygiene are the responsibility of the nurse. Patients on chemotherapy have risk for oral and systemic changes factors. The investigators will evaluate the cognitive and procedural knowledge about oral hygiene and the relevance of the learning experience importance.

DETAILED DESCRIPTION:
METHODOLOGY:

-Quasi-experimental research study, before and after an intervention, which was used in the educational video as a strategy for teaching about oral hygiene .

INSTRUMENTS:

1 ) tool to identify socio- demographic variables ( age, gender ),

2) scale (zero to ten) to assess the relevance of the student attaches the oral hygiene of people undergoing chemotherapy ;

3 ) instrument composed of true or false statements related to knowledge about oral hygiene for people undergoing chemotherapy,

4) instrument contemplating steps that should be used for oral hygiene of the patient and the structures escovadas6 ; contains a list of steps to observation record the implementation of the technique of brushing teeth , use mouthwash and floss;

5 ) rating scale the degree of acceptance of the use of video as educativa.7 the student carried out the technical strategy in itself ( before and after video ) , demonstrating how a patient undergoing chemotherapy should perform this technique .

The estimate for the subject's participation in research time was approximately 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

-Students in the fourth year of the Bachelor and the fifth year of undergraduate School of Nursing of Ribeirão Preto, University of São Paulo - USP

Exclusion Criteria:

-Desire to withdraw consent for the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Knowledge | In 30 minutes of the study (video and technique after and before that)
  * Effectiveness of an educational video on the cognitive and procedural knowledge of undergraduate students on the technique of oral hygiene in patients on chemotherapy;
  * Importance that the student attaches to this procedure for the oral health of people undergoing chemotherapy;
  * Acceptance of the use of a teaching strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Carvalho, Full professor, Principal Investigator — University of Sao Paulo
Locations (1):
- Escola de Enfermagem de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo, Brazil